CLINICAL TRIAL: NCT05651048
Title: The Role of BEMER and Kinesiotape in Increasing the Effectiveness of Physiotherapy and
Brief Title: The Role of BEMER and Kinesiotape in Increasing the Effectiveness of Physiotherapy and Rehabilitation Program After Videothoracoscopy Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, MAKBULE KARCI, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ICU-KARCI-3477
Record Dates: First submitted 2022-11-11; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Pain, Post Operative
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BEMER Group (Experimental): BEMER application with routine treatment protocol
  Interventions: Other: BEMER Group
- Kinesiotape Group (Experimental): Kinesiotape application with routine treatment protocol
  Interventions: Other: Kinesiotape Group
- Control Group (Experimental): routine treatment protocol
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Control Group — Physiotherapy and Rehabilitation Program After Videothoracoscopy Surgery
  Arms: Control Group
Other: BEMER Group — BEMER therapy and Physiotherapy and Rehabilitation Program After Videothoracoscopy Surgery
  Arms: BEMER Group
Other: Kinesiotape Group — Kinesiotape application and Physiotherapy and Rehabilitation Program After Videothoracoscopy Surgery
  Arms: Kinesiotape Group

SUMMARY:
The literature indicates that postoperative pulmonary complications are seen when pain is not treated effectively after videothoracoscopy surgery (VATS). After surgery, physiotherapy and rehabilitation approaches are applied to prevent complications. Bio-Electro-Magnetic-Energy-Regulation (BEMER) therapy uses low-frequency electromagnetic energy to regulate vasomotion in capillaries and increase microcirculation. BEMER therapy can be applied together with physiotherapy and rehabilitation. The aim of this study is to investigate the effectiveness of BEMER application, which is added to the physiotherapy and rehabilitation program applied after videothoracoscopy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study were to have undergone VATS lobectomy and to be aged between 18 and 75 years.

Exclusion Criteria:

* Presence of pacemaker, severe cardiac failure, severe arrhythmia
* Those with cooperative disorders
* Presence of neurological or orthopedic problems affecting the extremities
* Those with severe psychiatric disorders
* Failure to perform the operation according to the result of intraoperative tumor staging
* Patients who go out of the standard Analgesia protocol
* Patients who were taken back from the service to the intensive care unit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores | Postoperative 4th day
  Change From Baseline in Pain Scores on the Visual Analog Scale at Postoperative 4th day

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No